CLINICAL TRIAL: NCT01050452
Title: Gaps in Helminth Control: Safety and Efficacy of Drug Combinations. Study on Trichuris Trichiura.
Brief Title: Safety and Efficacy of Drug Combinations Against Trichuris Trichiura
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Responsible Party: Harriet Namwanje Principal Investigator, Vector control division, Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AO.UGA.TRI; DBL-CHRD
Record Dates: First submitted 2008-01-22; First posted 2010-01-15 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Parasitic Diseases
MeSH Terms: conditions — Parasitic Diseases | interventions — Albendazole; Mebendazole; Ivermectin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator): albendazole treatment
  Interventions: Drug: albendazole
- 2 (Active Comparator): mebendazole treatment
  Interventions: Drug: mebendazole
- 3 (Active Comparator): ivermectin treatment
  Interventions: Drug: ivermectin
- 4 (Active Comparator): albendazole + ivermectin treatment
  Interventions: Drug: albendazole + ivermectin
- 5 (Active Comparator): mebendazole + ivermectin treatment
  Interventions: Drug: mebendazole + ivermectin

INTERVENTIONS:
Drug: albendazole — albendazole (400 mg on dose)
  Arms: 1
Drug: mebendazole — mebendazole (500 mg one dose)
  Arms: 2
Drug: ivermectin — ivermectin (200 microgram/kg body weight)
  Arms: 3
Drug: albendazole + ivermectin — albendazole (400 mg one dose) + ivermectin (200 mg microgram/kg body weight)
  Arms: 4
Drug: mebendazole + ivermectin — mebendazole (500 mg one dose) + ivermectin (200 microgram/kg body weight)
  Arms: 5

SUMMARY:
This randomised, controlled, double-blinded clinical study investigates the safety and efficacy of albendazole (ALB), mebendazole (MBD) and ivermectin (IVM) separately, and ALB and MBD each in combination with IVM in the treatment of Trichuris trichiura in children aged 5-14 years.

ELIGIBILITY:
Inclusion Criteria:

* Those who are enrolled in class one to six
* Are infected with T. trichiura
* Whose parent consent and who are willing to participate

Exclusion Criteria:

* Those with acute and chronic diseases other than T. trichiura
* Those with a history of any serious adverse drug reactions

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 750 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Record adverse reactions | 6 weeks

SECONDARY OUTCOMES:
Efficacy of treatment | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Vector Control Division, Kampala, Uganda

REFERENCES:
- [Derived] Namwanje H, Kabatereine NB, Olsen A. Efficacy of single and double doses of albendazole and mebendazole alone and in combination in the treatment of Trichuris trichiura in school-age children in Uganda. Trans R Soc Trop Med Hyg. 2011 Oct;105(10):586-90. doi: 10.1016/j.trstmh.2011.07.009. Epub 2011 Aug 31. PMID 21885077